# **Informed Consent Form**

Effect of Different Neuromuscular Training Modalities on Postural Stability in Healthy Recreation People: A Randomised Controlled Trial

#### **Informed Consent Form**

TITLE OF STUDY: Effect of Different Neuromuscular Training Modalities on Postural

Stability in Healthy Recreation People: A Randomised Controlled Trial

Brief title: "Neuromuscular Training & Postural Stability"

**Acronym: STABLEFIT** 

#### PRINCIPAL INVESTIGATOR

Dragan Marinković

Faculty of sport and physical education University of Novi Sad, Srbia

# **PURPOSE OF STUDY**

Purpose of this study is to determine the effects of dynamic neuromuscular stabilization (DNS), whole-body vibration (WBV), and a combination of DNS and WBV (MIX) training modalities on postural stability (PS) in healthy recreation participants.

## STUDY PROCEDURES

Initial testing of postural stability on force platform as well as body weight, body height, age, gender.

Intervention (DNS, Vibration training, Mix of DNS and Vibration training; Control – no training)

Initial testing of postural stability on force platform

#### RISKS

No risk

#### **BENEFITS**

Improvement of postural stability and general health status.

#### **CONFIDENTIALITY**

For the purposes of this research study, your comments will not be anonymous. Every effort will be made by the researcher to preserve your confidentiality. Participant data will be kept confidential except in cases where the researcher is legally obligated to report specific incidents. These incidents include, but may not be limited to, incidents of abuse and suicide risk.

## **CONTACT INFORMATION**

If you have questions at any time about this study, or you experience adverse effects as the result of participating in this study, you may contact the researcher whose contact information is provided on the first page. If you have questions regarding your rights as a research participant, or if problems arise which you do not feel you can discuss with the Primary Investigator, please contact the Institutional Review Board at +381 21 450 188

# **VOLUNTARY PARTICIPATION**

Your participation in this study is voluntary. It is up to you to decide whether or not to take part in this study. If you decide to take part in this study, you will be asked to sign a consent form. After you sign the consent form, you are still free to withdraw at any time and without giving a reason. Withdrawing from this study will not affect the relationship you have, if any, with the researcher. If you withdraw from the study before data collection is completed, your data will be returned to you or destroyed.

#### **CONSENT**

I have read and I understand the provided information and have had the opportunity to ask questions. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving a reason and without cost. I understand that I will be given a copy of this consent form. I voluntarily agree to take part in this study.

| Participant's signature | Date |
|--------------------------|------|
| Investigator's signature | Date |
| investigator's signature | Datc |